CLINICAL TRIAL: NCT01908179
Title: Markers of Prognosis and Response to Therapy in Patients With Metastatic Brain Tumors Undergoing Stereotactic Radiosurgery (SRS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SRS - Mets
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Brain Tumor
Keywords: Sterotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This registry study will evaluate patients with metastatic brain tumors undergoing, or having undergone, stereotactic radiosurgery (SRS) at Swedish Medical Center. Clinical outcomes will be evaluated at the 3, 6 and 12-month time points. Clinical data, SRS treatment data, and imaging data (including anatomic and advanced imaging sequences obtained prior to and serially following SRS) will be archived in an online informatics platform, specifically a metastatic brain tumor registry known as the Comprehensive Neuro-oncology Data Repository for Metastatic Tumors (CONDR - Mets).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 yo) with a pathological diagnosis of metastatic brain cancer
* Participants must have >4 tumors felt to require stereotactic radiosurgery
* Karnofsky scale of > 70 at the time of initial treatment
* Age < 80

Exclusion Criteria:

* Karnofsky scale <70
* Age > 80
* Inability to undergo MR imaging studies

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic brain tumors undergoing, or have undergone, sterotactic radiosurgery (SRS)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Quantitative measures of overall tumor volume will be performed for each subject at the time of SRS | At the time of SRS
Quantitative measures of tumor number will be performed for each subject at the time of SRS | At the time of SRS
Overall survival will be measured for each subject (in weeks from SRS to death) | Post-SRS

SECONDARY OUTCOMES:
Measures of ADC, rCBV, MTT and ktrans will be performed for each treated tumor at treatment and at 6 months following SRS | 6 months post SRS
Time to progression (in weeks) will be measured for each treated tumor | Post-SRS
Diagnosis of progression or radiation necrosis (made on clinical reflection at study's end) will be determined for tumors where diagnosis is in question at 6 and 12 months after SRS | 12 months post-SRS

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States